CLINICAL TRIAL: NCT06868303
Title: A Quasi-controlled Study on the Effectiveness of Mental Wellness Youth Hubs in Hong Kong
Brief Title: The Effectiveness of Mental Wellness Youth Hubs in Hong Kong
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); The Boys' and Girls' Clubs Association of Hong Kong (Other); Caritas Medical Centre, Hong Kong (Other); Hong Kong Christian Service (Other); Neighbourhood Advice-Action Council (Other); St. James' Settlement (Other); Tung Wah Group of Hospitals (Other); Hong Kong Young Women's Christian Association (Other); Yan Oi Tong (Unknown); Chinese YMCA of Hong Kong (Unknown); New Life Psychiatric Rehabilitation Association (Other); The Salvation Army, Hong Kong and Macau Command (Other); Hong Kong Playground Association (HKPA) (Unknown); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Hong Kong Children and Youth Services (HKCYS) (Unknown); Hong Kong Federation of Youth's Group (HKFYG) (Other)
Responsible Party: Principal Investigator, Dr. Christy Lai-ming Hui, Associate Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250221-005-000
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Mental Stress
Keywords: Youth Mental Health
MeSH Terms: conditions — Stress, Psychological | interventions — General Practitioners

STUDY DESIGN:
Intervention Model Description: The experiment group will include 600 hub users who are not currently using psychiatric medications and do not have a formal diagnosis at the time of enrolling in the hub activity. The control group will also comprise of 600 young people, recruited from a community cohort managed by the research team. For the substudy examining the impact of the service model, a total of 252 participants will be recruited, with 63 individuals selected from each of the following groups: those receiving services through NLPRA eClinic, accessing care via the Integrated Community Centre for Mental Wellness (ICCMW) step-up program, managed by general practitioners, and isupported by hub casework services. For the substudy evaluating the impact pf Tier 1 activities, young people experiencing Tier 1 distress levels (determined by K6 < 11), who have participated only in Tier 1 activities, will be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Hub User Group (Experimental): This group receives community-based mental wellness youth hub services for young people to enhance personal strengths and overall mental well-being.
  Interventions: Behavioral: LevelMind@JC Mental Wellness Youth Hubs
- Non-hub User Community Control Group (No Intervention): This group does not receive any youth services in the community.
- eClinic User Group (Active Comparator): This group receives the eClinic service provided by New Life Psychiatric Rehabilitation Association.
  Interventions: Behavioral: New Life Psychiatric Rehabilitation Association electronic clinic for psychological service
- ICCMW group (Active Comparator): This group receives the eClinic service provided by Integrated Community Centre for Mental Wellness (ICCMW) step-up care.
  Interventions: Behavioral: Integrated Community Centres for Mental Wellness
- GP group (Active Comparator): This group receives services provided by general practitioners.
  Interventions: Other: General Practitioner
- Hub Casework grpup (Active Comparator): This group receives services from hub casework support, as well as from NLPRA eClinic, ICCMW, and general practitioners.
  Interventions: Behavioral: New Life Psychiatric Rehabilitation Association electronic clinic for psychological service; Behavioral: Integrated Community Centres for Mental Wellness; Other: General Practitioner; Behavioral: Hub Casework

INTERVENTIONS:
Behavioral: LevelMind@JC Mental Wellness Youth Hubs — Mental Wellness Youth Hubs Intervention aims to set up a series of community-based hubs for young people to enhance cognitive abilities, personal strengths and overall mental well-being. Among the experimental group participants (hub users), they are further divided into three tiers according to their psychological distress level. Tier 1 are youths with mild psychological distress level, who will be invited to participate in some innovative and interesting youth projects and activities (e.g., board game and floral artistry). Tier 2 are youths who have moderate level of psychological distress, or at risk for mental illness. Trained social workers will offer them with specific interventions (e.g., CBT, sleep intervention) according to their needs. Tier 3 are youths with severe level of psychological distress who are at risk for mental disorders. Diagnostic and medical assessment services will be delivered by psychiatrist or clinical psychologists.
  Arms: Hub User Group
Behavioral: New Life Psychiatric Rehabilitation Association electronic clinic for psychological service — The eClinic treatment spans eight to fourteen week and is designed for individuals with moderate to severe mental health issues. The service is provided in a hybrid format, incorporating an in-person initial screening using the Patient Health Questionnaire-9 and General Anxiety Disorder-7, followed by online self-learning resources and sessions with a therapist. Pre- and post-treatment assessments as well as follow-ups will be used to keep track of service users' progress.
  Arms: Hub Casework grpup; eClinic User Group
Behavioral: Integrated Community Centres for Mental Wellness — Integrated Community Centres for Mental Wellness (ICCMWs) are the main community-based mental health services in Hong Kong. However, their reach among young people is limited, as their broad target age range primarily focuses on middle-aged individuals. ICCMW offers comprehensive, district-based community support and social rehabilitation services, from early prevention to risk management, for people in mental recovery, those with suspected mental health issues, their families and carers, and residents within the service area, all accessible through a single-entry point.
  Arms: Hub Casework grpup; ICCMW group
Other: General Practitioner — Services provided by genersl practitioner
  Arms: GP group; Hub Casework grpup
Behavioral: Hub Casework — Services provided during hub casework sessions
  Arms: Hub Casework grpup

SUMMARY:
This study sets out to evaluate (i) whether the model in phase two can improve symptoms, quality of life, functioning, and psychological outcomes in young people utilising the hub services (n = 600) compared to those in the community controls (n = 600), (ii) the mechanisms that may drive these improvements, and (iii) whether any particular subgroup(s) of youths (e.g., gender, socio-economic status, migrant status) may benefit more from this service model. The experiment group will include 600 hub users who are not currently using psychiatric medications and do not have a formal diagnosis at the time of enrolling in the hub activity. The control group will also comprise of 600 young people, recruited from a community cohort managed by the research team. The community cohort is accessible via the Youth Epidemiological Study Online platform (YES online), which recruits young people aged 12 to 24 years. Only YES online participants who are not using the service of LevelMind@JC and psychiatric medications will be recruited for this study. The two groups will be matched in age, gender, and baseline distress level measured by the 6-item Kessler Psychological Distress Scale (K6). There will also be a substudy assessing the effect of four service models: NLPRA eClinic, Integrated Community Centre for Mental Wellness (ICCMW) step-up care, general practitioners, and hub casework support service on symptom-based mental health outcome, comparing a cohort of young people receiving these four services respectively. A total of 252 participants will be recrruited. Another substudy will be conducted to investigate the extent to which participation in Tier 1 activities contributes to improvements in targeted outcome areas, assessing young people (n = 675) before and after their participation of Tier 1 activities. A consecutive sampling will be used, where a subject who meets the criteria of inclusion will be selected until this required sample size is achieved.

ELIGIBILITY:
Inclusion Criteria:

* For hub user group: 12- to 24-year-old hub users who receive community-based mental wellness youth hub services for young people.
* For community control group: 12- to 24-year-old community youths who do not receive any youth services in the community.
* For eClinic user group: 12- to 24-year-old eClinic service users.

Exclusion Criteria:

* Youths with known diagnosis of psychiatric disorders (including Depression, Generalized Anxiety Disorder, Panic Disorder, Phobia, Obsessive Compulsive Disorder, Bipolar Disorder, Eating Disorder, Personality Disorder, Post-Traumatic Stress Disorder and Psychotic Disorder)
* Youths who receive psychiatric medication (including antidepressants, antipsychotics and antiepileptic drugs)

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Distress | Baseline, 3-month, 6-month, and 12-month
  The 6-item Kessler Psychological Distress Scale (scores range from 0 to 24 where a higher score indicates a worse outcome)
Change in Well-being | Baseline, 3-month, 6-month, and 12-month
  The World Health Organization-Five Well-Being Index (scores range from 0 to 25 where a higher score indicates a better outcome)
Change in Quality of Life | Baseline, 3-month, 6-month, and 12-month
  The 12-item Short-Form 12 Health Survey (scores range from 0 to 100 where a higher score indicates a better outcome)

SECONDARY OUTCOMES:
Change in Depressive, Anxiety, and Stress Levels | Baseline, 3-month, 6-month, and 12-month
  The 21-item Depression Anxiety Stress Scales (scores range from 0 to 63 where a higher score indicates a worse outcome)
Change in Social and Occupational Functioning | Baseline, 3-month, 6-month, and 12-month
  Social and Occupational Functioning Assessment Scale (scores range from 0 to 100 where a higher score indicates a better outcome)
Change in Sleep Quality | Baseline, 3-month, 6-month, and 12-month
  Pittsburgh Sleep Quality Index (scores range from 0 to 21 where a higher score indicates a worse outcome)
Change in Physical Exercise | Baseline, 3-month, 6-month, and 12-month
  The International Physical Activity Questionnaire (classify physical activity level into three categories: low, moderate, and high)
Change in Self-Esteem Level | Baseline, 3-month, 6-month, and 12-month
  Rosenberg Self-Esteem Scale (scores range from 0 to 30 where a higher score indicates a better outcome)
Change in Psychological Resilience | Baseline, 3-month, 6-month, and 12-month
  The 10-item Connor-Davidson Resilience Scale (scores range from 0 to 40 where a higher score indicates a better outcome)
Change in Cognitive Function | Baseline, 3-month, 6-month, and 12-month
  Digit Span Test
Change in Health Economics | Baseline, 3-month, 6-month, and 12-month
  Client Service Receipt Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Christy Lai Ming Hui, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Community, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No